CLINICAL TRIAL: NCT03602612
Title: A Phase I Clinical Trial of T Cells Expressing a Novel Fully-human Anti-BCMA CAR for Treating Multiple Myeloma
Brief Title: T Cells Expressing a Novel Fully-Human Anti-BCMA CAR for Treating Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Kochenderfer, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180125; 18-C-0125
Record Dates: First submitted 2018-07-26; First posted 2018-07-27 (Actual); Results first posted 2023-05-15 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Myeloma-Multiple; Myeloma, Plasma-Cell
Keywords: B-cell Maturation Antigen; Immunotherapy; Chimeric Antigen Receptors; Adoptive T Cell Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; bis(3-bis(4-chlorophenyl)methyl-4-dimethylaminophenyl)amine; Receptors, Chimeric Antigen; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Conditioning chemotherapy plus chimeric antigen receptors (CARs) T-cells dose escalation (Experimental): Patients will receive escalating doses (up to 5 planned) of CAR+ T cells infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Anti-B Cell Maturation Antigen (BCMA) chimeric antigen receptors (CARs) T cells
- 2/Conditioning chemotherapy plus chimeric antigen receptors (CARs) T-cells expansion phase (Experimental): 6.0x10^6 dose (maximum feasible dose) of CAR T Cells + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Anti-B Cell Maturation Antigen (BCMA) chimeric antigen receptors (CARs) T cells

INTERVENTIONS:
Drug: Cyclophosphamide — 300 mg/m^2 intravenous (IV) over 30 minutes on days -5, -4, and -3
  Other Names: Cytoxan
Drug: Fludarabine — 30 mg/m^2 intravenous (IV) infusion over 30 minutes administered immediately following the cyclophosphamide on day -5, -4, -3
  Other Names: Fludara
Biological: Anti-B Cell Maturation Antigen (BCMA) chimeric antigen receptors (CARs) T cells — 0.75x10^6 - 12.0X10^6 CAR+ T cells per kg of recipient bodyweight one time dose on day 0

SUMMARY:
Background:

Multiple myeloma is a cancer of the blood plasma cells. It usually becomes resistant to standard treatments. Researchers have developed a procedure called gene therapy. It uses a person's own T cells, which are part of the immune system. The cells are changed in a lab and then returned to the person. Researchers hope the changed T cells will be better at recognizing and killing tumor cells.

Objective:

To test the safety of giving changed T cells to people with multiple myeloma.

Eligibility:

Adults ages 18-73 who have been diagnosed with multiple myeloma that has not been controlled with standard therapies.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood tests

Heart function tests

Bone marrow sample taken by needle in a hip bone.

Scan of the chest, abdomen, and pelvis. They may have a brain scan.

Pregnancy test

Participants will have apheresis. Blood will be removed through an arm vein. The blood will be separated, and T cells removed. The rest of the blood will be returned through a vein in the other arm.

Participants will have a central line placed in a large vein in the arm or chest.

Participants will get 2 chemotherapy drugs by the central line over 3 days.

Two days later, participants will get the changed T cells by the central line. They will stay in the hospital at least 9 days.

Participants must stay near the hospital for 2 weeks.

Participants will have 8 follow-up visits over the next year for blood and urine tests. They may have scans.

Participants blood will be collected regularly over the next several years.

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is a malignancy of plasma cells.
* MM is nearly always incurable.
* T cells can be genetically modified to express chimeric antigen receptors (CARs) that specifically target malignancy-associated antigens.
* Autologous T cells genetically modified to express CARs targeting the B-cell antigen B-lymphocyte antigen CD19 (CD19) have caused complete remissions in a small number of patients with leukemia or lymphoma. These results demonstrate that CAR-expressing T cells have anti-malignancy activity in humans.
* B-cell maturation antigen (BCMA) is a protein expressed by normal plasma cells and the malignant plasma cells of multiple myeloma.
* BCMA is not expressed by normal cells except for plasma cells and some mature B cells.
* We have constructed a novel anti-BCMA CAR that can specifically recognize BCMA- expressing target cells in vitro and eradicate BCMA-expressing tumors in mice.
* This CAR has an antigen-recognition domain made up of a single fully-human heavy chain variable region.
* We hypothesize that anti-BCMA-CAR-expressing T cells will specifically eliminate BCMA- expressing MM cells in patients
* Possible toxicities include cytokine-associated toxicities such as fever, hypotension, and neurological toxicities. Elimination of normal plasma cells and unknown toxicities are also possible.

Objectives:

Primary

- Determine the safety and feasibility of administering T cells expressing an anti-BCMA CAR to patients with MM.

Eligibility:

* Greater than or equal to 18 years of age and less than or equal to age 73.
* Patients must have measurable MM defined as a serum M-protein greater than or equal to 1.0 g/dL or a urine M- protein greater than or equal to 200 mg/24 hours or an involved serum free light chain (FLC) level greater than or equal to 10 mg/dL (provided FLC ratio is abnormal) or a biopsy-proven plasmacytoma of 2.0 cm or more in largest dimension, or greater than or equal to 30% bone marrow plasma cells
* Patients must have previously received at least 3 different treatment regimens for MM.
* Patients must have prior exposure to an immunomodulatory imide drugs (IMiD) such as lenalidomide, and a proteasome inhibitor
* Patients must have a creatinine level of less than or equal to 1.5 mg/dL
* Patients must have a cardiac ejection fraction greater than or equal to 50%.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 is required.
* Patients on any anticoagulant medications except aspirin are not eligible.
* No active infections are allowed.
* Absolute neutrophil count greater than or equal to 1000/microliters, platelet count greater than or equal to 55,000/ microliters, hemoglobin greater than or equal to 8g/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5-fold higher than the upper limit of normal.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and the required leukapheresis.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and initiation of protocol treatment.
* The patients MM will need to be assessed for BCMA expression by flow cytometry or immunohistochemistry performed at the National Institutes of Health (NIH). The myeloma must express BCMA. If unstained, paraffin-embedded bone marrow or plasmacytoma sections are available from prior biopsies, these can be used to determine BCMA expression by immunohistochemistry; otherwise, patients will need to come to the NIH for a bone marrow biopsy or other biopsy of a plasmacytoma to determine BCMA expression. The sample for BCMA expression can come from a biopsy obtained at any time before enrollment.

Design:

* This is a phase I dose-escalation trial
* Patients will undergo leukapheresis
* T-cells obtained by leukapheresis will be genetically modified to express an anti-BCMA CAR
* Patients will receive a lymphocyte-depleting chemotherapy conditioning regimen with the intent of enhancing the activity of the infused anti-BCMA-CAR-expressing T cells.
* The chemotherapy conditioning regimen is cyclophosphamide 300 mg/m^2 daily for 3 days and fludarabine 30 mg/m^2 daily for 3 days. Fludarabine will be given on the same days as the cyclophosphamide.
* After the chemotherapy ends, the patients will have two days with no treatments then receive an infusion of anti-BCMA- CAR-expressing T cells.
* The initial dose level will be 0.75x10^6 CAR+ T cells/kg of recipient bodyweight.
* The cell dose administered will be escalated until a maximum tolerated dose is determined.
* Following the T-cell infusion there will be a mandatory 9-day minimum inpatient hospitalization to monitor for toxicity.
* Outpatient follow-up is planned for 2 weeks, and 1, 2, 3, 4, 6, 9, and 12 months after the CAR T-cell infusion. Afterwards, follow-up will be every six months up to at least 5 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

Multiple Myeloma (MM) criteria:

* B Cell Maturation Antigen (BCMA) expression must be detected on malignant plasma cells from either bone marrow or a plasmacytoma by flow cytometry or immunohistochemistry. If patient has plasmacytomas, one plasmacytoma must be biopsied to demonstrate BCMA expression. A specific quantitative level of BCMA expression for eligibility is not specified, but patients with multiple myeloma cells that are negative for BCMA by flow cytometry and immunohistochemistry on either bone marrow biopsy or plasmacytoma biopsy will not be enrolled. These assays must be performed at the National Institutes of Health (NIH). It is not required that the specimen used for BCMA determination comes from a sample that was obtained after the patients most recent treatment. If paraffin embedded unstained samples of bone marrow involved with MM or a plasmacytoma are available, these can be shipped to the NIH for BCMA staining, otherwise new biopsies will need to be performed for determination of BCMA expression.
* BCMA expression will need to be documented on the majority of malignant plasma cells by flow cytometry at the NIH at some time after the original anti-BCMA chimeric antigen receptors (CARs) T-cell infusion in all patients undergoing a second anti-BCMA CAR T-cell infusion.
* Bone marrow plasma cells must make up less than 50% of total bone marrow cells based on a bone marrow biopsy performed within 24 days of the start of protocol treatment.
* Patients must have received at least 3 different prior treatment regimens for multiple myeloma
* Must have prior exposure to an immunomodulatory imide drugs ("IMiD") such as lenalidamide and a proteasome inhibitor
* Patients must have measurable MM as defined by at least one of the criteria below.

  * One or more of these abnormalities defines measurable multiple myeloma:
  * Serum M-protein greater or equal to 1.0 g/dL.
  * Urine M-protein greater or equal to 200 mg/24 h.
  * Serum free light chain (FLC) assay: involved FLC level greater or equal to 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal.
  * A biopsy-proven plasmacytoma at least 2.0 cm in largest dimension
  * Bone marrow core biopsy with 30% or more plasma cells

Other inclusion criteria:

* Greater than or equal to 18 years of age and less than or equal to age 73.
* Able to understand and sign the Informed Consent Document.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-2
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after last day of receiving protocol treatment.
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
* A patient with a negative blood polymerase chain reaction (PCR) test for hepatitis B deoxyribonucleic acid (DNA) test can be enrolled. If hepatitis B DNA (PCR) testing is not available, patients with a negative hepatitis B surface antigen and negative hepatitis B core antibody can be enrolled.
* Patients must be tested for the presence of Hepatitis C antigen by PCR and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative in order to be eligible. Only if Hepatitis C PCR testing is not available in a timely manner, patients who are Hepatitis C antibody-negative can be enrolled.
* Absolute neutrophil count greater than or equal to 1000/mm(3) without the support of filgrastim or other growth factors within the previous 10 days.
* Platelet count greater than or equal to 55,000/mm(3) without transfusion support within the past 10 days.
* Hemoglobin greater than 8.0 g/dL
* Less than 5% plasma cells in the peripheral blood leukocytes
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of the institutional normal.
* Serum creatinine less than or equal to 1.5 mg/dL.
* Total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilberts Syndrome who must have a total bilirubin less than 3.0 mg/dL.
* At least 14 days must have elapsed since any prior systemic therapy at the time the patient starts the cyclophosphamide and fludarabine conditioning regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
* Because this protocol requires collection of autologous blood cells by leukapheresis in order to prepare anti-BCMA-CAR T cells, systemic anti-myeloma therapy including systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 2 weeks prior to the required leukapheresis.
* Normal cardiac ejection fraction (greater than or equal to 50% by echocardiography) and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram.
* For patients with past participation in gene-therapy, cryopreserved peripheral blood mononuclear cells (PBMCs) that have not been genetically engineered must be available.

EXCLUSION CRITERIA:

* Patients on any anticoagulants except aspirin.
* Patients that require urgent therapy due to tumor mass effects or spinal cord compression.
* Patients that have active hemolytic anemia.
* Patients with second malignancies in addition to multiple myeloma are not eligible if the second malignancy has required treatment within the past 3 years or is not in complete remission. There are two exceptions to this criterion: successfully treated non-metastatic basal cell or squamous cell skin carcinoma.
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Women of child-bearing potential cannot have a positive pregnancy test. Women of child-bearing potential are defined as all women except women who are post-menopausal or who have had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
* Active systemic infections (defined as infections causing fevers or requiring anti- microbial treatment), active coagulation disorders or other major uncontrolled medical illnesses of the cardiovascular, respiratory, endocrine, renal, gastrointestinal, genitourinary, neurologic, or immune system, history of myocardial infarction, active cardiac arrhythmias including active atrial fibrillation history of any arrhythmias other than sinus tachycardia, or atrial fibrillation, currently taking any anti-arrythmic or congestive heart failure medications, active obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid (prednisone, dexamethasone, etc.) is not allowed within 2 weeks prior to either the required leukapheresis or within 2 weeks prior to CAR T-cell infusion (and at any time after the CAR T cell infusion).
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Patient unwilling to undergo intensive care unit treatment including mechanical ventilation, cardiopulmonary resuscitation, vasoactive drugs, and hemodialysis.
* History of allogeneic stem cell transplantation
* Patients with current spinal cord compression (without intradural myeloma involvement).
* Patients who have a history (or current evidence) of cerebrospinal fluid multiple myeloma, or intra-dural central nervous system masse
* Patients with active autoimmune skin diseases such as psoriasis or other active autoimmune diseases such as rheumatoid arthritis.
* Patients must not have required supplemental oxygen within the past month unless it was for a resolved infection.
* Patient must not have received genetically modified cells except on prior National Cancer Institute (NCI) gene therapy protocols.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2026-04-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0125.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Dose Escalation Dose Level (DL) -1 - 0.4x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg: Participants received 0.4x10^6 Chimeric Antigen Receptor (CAR)+ T cells per kg infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3.
- Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg: Participants received 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T cells per kg infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3.
- Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg: Participants received 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T cells per kg infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3.
- Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg: Participants received 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T cells per kg infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3.
- Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg: Participants received 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T cells per kg infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3.
- Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg: Participants received 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T cells per kg infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3.
- Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg: Participants received 6.0x10^6 (maximum feasible dose) CAR+T cells per kg + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg: Dose Escalation: Participants received 3.0x10^6 CAR+T cells per kg infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3.
  AND
  Dose Expansion:
  Participants received 6.0x10^6 (maximum feasible dose) CAR+T cells per kg + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
- Participants Enrolled in Arm 1 But Not Treated; Participants Enrolled in Arm 2 But Not Treated: Participants was enrolled but not treated.
Period: Dose Escalation Phase
Arm/Group | Arm 1 Dose Escalation Dose Level (DL) -1 - 0.4x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg | Participants Enrolled in Arm 1 But Not Treated | Participants Enrolled in Arm 2 But Not Treated
Started | 0 (No participants were enrolled in this Arm/Group.) | 6 | 3 | 2 | 3 | 3 | 0 | 1 | 8 | 1
Completed | 0 | 6 | 3 | 2 | 3 | 3 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 1
Period: Dose Expansion Phase
Arm/Group | Arm 1 Dose Escalation Dose Level (DL) -1 - 0.4x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg | Participants Enrolled in Arm 1 But Not Treated | Participants Enrolled in Arm 2 But Not Treated
Started | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data collected for two participants enrolled but not treated is reported here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg | Participants Enrolled in Arm 1 But Not Treated | Participants Enrolled in Arm 2 But Not Treated | Total
Number analyzed (Participants) | 6 | 3 | 2 | 3 | 3 | 8 | 1 | 8 | 1 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 1 | 1 | 2 | 5 | 1 | 6 | 1 | 23
  >=65 years | 3 | 0 | 1 | 2 | 1 | 3 | 0 | 2 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.57 (13.26) | 57.47 (5.59) | 61.6 (12.59) | 62.63 (9.79) | 56.57 (8.48) | 62.03 (9.41) | 64.4 (0) | 54.86 (10.11) | 50.9 (0) | 58.54 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 1 | 5 | 1 | 5 | 0 | 20
  Male | 4 | 1 | 0 | 1 | 2 | 3 | 0 | 3 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 2 | 1 | 3 | 3 | 7 | 1 | 7 | 1 | 29
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 10
  White | 1 | 0 | 2 | 2 | 2 | 6 | 1 | 3 | 1 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 2 | 3 | 3 | 8 | 1 | 8 | 1 | 35

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Anti-B Cell Maturation Antigen (BCMA) - Chimeric Antigen Receptor (CAR)-T Cells
Description: The MTD is the dose at which a maximum of 1 of 6 patients has a DLT. A DLT is Grade 3 toxicities possibly or probably or definitely related to the Anti-B cell maturation antigen (BCMA) - chimeric antigen receptor (CAR)-expressing T-Cells lasting more than 9 days. Grade 4 toxicities possibly or probably or definitely related to the anti-BCMA CAR T cells. Grade 3 is severe, and Grade 4 is life-threatening.
Time Frame: First 28 days of treatment
Population: 9/35 participants were enrolled but not treated.
Measure: Number; unit: million CAR + T cells
Groups:
- All Arm 1 Dose Escalation Dose Participants: All participants in Arm 1 Dose Escalation Group who received CAR+T cells, Cyclophosphamide and Fludarabine.
Arm/Group | All Arm 1 Dose Escalation Dose Participants
Number analyzed (Participants) | 18
million CAR + T cells | 6

2. Primary Outcome: Number of Participants at Each Dose Level Who Experience a Dose-Limiting Toxicity (DLT)
Description: A DLT is Grade 3 toxicities possibly or probably or definitely related to the anti-B cell maturation antigen (BCMA) - chimeric antigen receptor (CAR)-T cells and lasting more than 9 days. Grade 4 toxicities possibly or probably or definitely related to the anti-BCMA CAR T cells. Grade 3 is severe, and Grade 4 is life-threatening.
Time Frame: First 28 days of treatment
Population: 9/35 participants were enrolled but not treated.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg: Dose Escalation: Participants received 3.0x10^6 CAR+T cells per kg infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg /m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3 AND Dose Expansion: Participants received 6.0x10^6 (maximum feasible dose) CAR+T cells per kg + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
Arm/Group | Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg
Number analyzed (Participants) | 6 | 3 | 2 | 3 | 3 | 8 | 1
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 16 months/17 days, 4 months/4 days, 4 months/18 days, 42 months/8 days, 20 months/19 days, 29 months/28 days, and 30 months/26 days for each Arm/Group respectively.
Population: 9/35 participants were enrolled but not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg
Number analyzed (Participants) | 6 | 3 | 2 | 3 | 3 | 8 | 1
Participants | 6 | 3 | 2 | 3 | 3 | 8 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 16 months/17 days, 4 months/4 days, 4 months/18 days, 42 months/8 days, 20 months/19 days, 29 months/28 days, and 30 months/26 days for each Arm/Group respectively.
Arm/Group | Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg | Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/3 | 0/2 | 0/3 | 0/3 | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 6/6 | 1/3 | 2/2 | 2/3 | 3/3 | 6/8 | 1/1
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 2/2 | 3/3 | 3/3 | 8/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=6) | Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=3) | Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=2) | Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=3) | Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=3) | Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=8) | Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nervous system disorders - Other, Saddle anesthesia with pinprick below the mid calves. (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure - death (due to influenza) grade 5 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon reflex decreased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Dose Escalation (Esc) Dose Level 1 - 0.75x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=6) | Arm 1 Dose Escalation Dose Level 2 - 1.5x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=3) | Arm 1 Dose Escalation Dose Level 3 - 3.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=2) | Arm 1 Dose Escalation Dose Level 4 - 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=3) | Arm 1 Dose Escalation Dose Level 5 - 12.0x1^06 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=3) | Arm 2 Dose Expansion (Exp) 6.0x10^6 Chimeric Antigen Receptor (CAR)+ T Cells Per kg (N=8) | Arm 1 DoseEsc DL 3-3.0x10^6 CAR+T Cells Per kg Followed by Arm 2 DoseExp 6.0x10^6 CAR+T Cells Per kg (N=1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 6 (47) | 3 (12) | 2 (11) | 2 (15) | 3 (22) | 8 (48) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (5) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CPK increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (6) | 1 (1) | 1 (1) | 5 (11) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, new diagnosis of Fuchs corneal dystrophy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 6 (13) | 0 (0)
Fever (General disorders) | 5 (7) | 2 (2) | 2 (3) | 3 (4) | 3 (12) | 7 (14) | 1 (4)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal disorders - Other, Bilateral hernias (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, Fatty liver (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (14) | 1 (1) | 1 (2) | 1 (3) | 2 (9) | 5 (17) | 1 (8)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (10) | 1 (1) | 1 (5) | 3 (3) | 3 (8) | 6 (10) | 1 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (12) | 0 (0) | 2 (5) | 2 (3) | 3 (6) | 5 (15) | 1 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (18) | 1 (2) | 2 (5) | 2 (10) | 3 (9) | 7 (24) | 1 (4)
Hypotension (Vascular disorders) | 2 (2) | 2 (6) | 1 (1) | 1 (2) | 1 (1) | 5 (6) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Staph capitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Two ticks found on right thigh on 7/20/19, and were removed. (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, cough and chest congestion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, fevers, fatigue, URI symptoms (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Investigations - Other, B12 low normal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, Specify (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Vit D Deficiency 20 ng/mL, weekly high dose vitamin D for 8 weeks (started 12/31)
Investigations - Other, Vit D deficiency 24 ng/mL (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (35) | 3 (12) | 1 (5) | 3 (19) | 3 (22) | 8 (33) | 1 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 5 (6) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Squamous cell carcinoma, LUE
Nervous system disorders - Other, Decreased sensation L>R LE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, Diffuse loss of fine touch sensation over the mid-abdomen (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (50) | 3 (22) | 2 (17) | 3 (14) | 3 (23) | 8 (80) | 1 (14)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 3 (17) | 1 (9) | 2 (11) | 2 (13) | 3 (12) | 7 (34) | 1 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Repiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 7 (8) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, actinic keratoses (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Cataract surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (8) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 6 (59) | 3 (32) | 2 (15) | 3 (18) | 3 (25) | 8 (95) | 1 (16)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, Earlobe trauma (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Restless Leg Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of the jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03602612/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT03602612/ICF_002.pdf